CLINICAL TRIAL: NCT04337814
Title: The Effect of Combined Oral and Topical Analgesics to Reduce Pain Perception During Electromyography in Pediatric Population-A Randomized Controlled Trial
Brief Title: The Effect of Combined Oral and Topical Analgesics to Reduce Pain Perception During Electrodiagnostic Testing
Acronym: COMFORTEMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Fazal ur Rehman, Principal Inestigator, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2019-0631-4863
Record Dates: First submitted 2019-12-16; First posted 2020-04-08 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Pain Perception
Keywords: Electromyopharpy; Nerve conduction study; Electrodiagnostic testing; Edx study; EMG; NCS
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled randamized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- COTA Arm (Experimental): Patients getting combined (C) oral (O) and topical (T) analgesics (A)
  Interventions: Drug: EMLA Cream; Drug: Ibuprofen
- OA Arm (Experimental): Patients getting oral (O) analgesics (A) and topical placebo
  Interventions: Drug: Ibuprofen; Drug: Placebo cream
- Placebo Arm (Placebo Comparator): Patients getting oral placebo and topical placebo
  Interventions: Drug: Placebo syrup; Drug: Placebo cream

INTERVENTIONS:
Drug: EMLA Cream — Topical anaesthetic cream
  Arms: COTA Arm
Drug: Ibuprofen — Oral analgesic syrup (non-steroidal anti inflammatory drug)
  Arms: COTA Arm; OA Arm
Drug: Placebo syrup — Placebo syrup similar to Ibuprofen
  Arms: Placebo Arm
Drug: Placebo cream — Placebo cream similar to EMLA
  Arms: OA Arm; Placebo Arm

SUMMARY:
Electromyography (EMG) is a useful test for diagnosis and monitoring of lower motor neuron disorders. It is mostly done in conjunction with a Nerve Conduction Study (NCS). Like other invasive medical procedures; electrodiagnostic tests have been known to cause iatrogenic pain for the patient, the intensity of which varies from person to person. Multiple modifiable as well as non-modifiable risk factors associated with EMG pain have been described in literature.Various approaches targeting different mechanisms of pain perception have been tested to make this procedure comfortable for the patients. These approaches range from simple distraction techniques to the use of topical and oral analgesics.Most of these studies have looked at adult population which has, supposedly, better pain tolerance as compared to children. Data on EMG associated pain in pediatric population is scant. This trial will assess the effect of combined oral and topical analgesics to reduce pain perception during NCS and EMG tests in the pediatric population.

DETAILED DESCRIPTION:
Objectives:

To determine the effect of combined oral and topical analgesics (COTA) in reducing pain perception during NCS and EMG tests among the pediatric population.

To compare the effect of COTA and only oral analgesics (OA) in reducing pain perception during NCS and EMG tests among the pediatric population.

Methods:

Study Setting: This study will be conducted at the neurophysiology lab at Aga Khan University Hospital (AKUH)

Study Design: This will be a stratified (6 months - 6 years and 7 - 18 years with balanced randomization), double-blind, placebo-controlled, parallel group study conducted at the neurophysiology lab, AKUH.

Variables:

Independent Variables - Gender, age, weight (Kg), number of muscles sampled, distribution of muscles sampled, end plate noise detection, type of needle used, duration of EMG and NCS test, history of undergoing electrodiagnostic tests in the past, time duration between analgesic intake / application and start of the NCS and EMG test, number of needle insertions needed outside of applied cream area, number of times skin is pierced,result of electrodiagnostic examination, patient in parents lap, electromyographer, study arm.

Dependent Variables - Pain Scores (MBPS and FPS-R)

Interventions/Study Protocol:

The guardians / patients who meet the inclusion criteria, as determined by the neurophysiology fellow or attending, will be instructed to reach the neurophysiology lab on the day of appointment one hour before the expected procedure time. All patients and/or their guardians referred for NCS / EMG will be given a standard explanation regarding the procedure and study details on the day of electrodiagnostic testing by the designated neurophysiology technologist. NCS would be explained as a test that checks the responses of the nerves and the subject will feel small zaps during the procedure. EMG would be explained as a procedure where a thin small microphone will be inserted in multiple muscles of the arm, leg and / or neck and back that will help us in identifying the problem. The word 'needle' and 'electric current' would not be used during this explanation. The guardian and patient, if old enough to understand, will also be explained the study protocol being carried out. Written Informed consent for the procedure itself and the study will be taken at this point by the neurophysiology fellow. Patients (older than 6 years) or their guardians will be instructed on how to administer the FPS-R scale. In addition guardians would be instructed to make sure that patients are not given sugary drinks or breastfeed during 1 hour prior to the procedure. During the study distractions will be kept to a minimum and similar for all patients. Sites of needle insertion will not be rubbed, stroked or tapped at the time of needle insertion. These factors are known confounders in reducing intramuscular injection pain. Those who have given consent will be assigned to one of the three arms of the study according to the randomization schedule; COTA arm (Ibuprofen Syrup and EMLA Cream), OA arm (Ibuprofen Syrup and Plain Cream) or Placebo arm (Plain Syrup and Plain Cream). All patients will be issued their interventions labeled with an allocation sequence according to the randomization schedule from the clinical trials unit (CTU), in a double blind manner, on the day of appointment. The syrup will be given to patients orally (10mg/Kg body weight) at least 1 hour prior to start of procedure. The electromyographer will demarcate all the possible muscle sampling sites required as per study protocol with a non-toxic marker and leave the room. A neurophysiology technologist will apply the cream on all demarcated sites. After application of cream, the site would be covered by an occlusive dressing until NCS / EMG is carried out so as to keep the applied cream in place and prevent accidental ingestion or application on mucosal surfaces by the patient. The patient will be kept under observation for adverse reactions including blanching and local erythema from application of cream till 15 minutes after the NCS / EMG procedure. Observation would be done by Neurophysiology fellow or the Neurophysiology attending. Neurophysiology technologists designated to carry out this exercise would be given combined sessions regarding the application technique to achieve consistency in results.

The EMG will be performed by board certified faculty or neurophysiology fellows under their supervision, each of them having a minimum of 6 months experience in doing electrodiagnostic testing. This involves intramuscular insertion of needle (that has a microphone at its tip) into multiple muscles. The occlusive dressing will be removed and area to be tested wiped with alcohol swabs. Nerve conduction studies will be conducted first followed by the needle procedures. During nerve conduction studies, patients feel an electric current like sensation whenever a nerve is tested. Attempt will be made to keep the needle movements to minimum. The guardian would accompany the child throughout the procedure. If the child wants, he/she would be allowed to sit in the guardians lap during the procedure.

Pain Assessment & Data Collection:

For children aged 6 months to 6 years pain will be assessed by scoring facial expression, cry and body movements of the children using the Modified Behavioral Pain Scale (MBPS). For children aged 7 years to 18 years the Face Pain Scale-Revised (FPS-R) version will be used. Patients will be scored before NCS, after NCS and after EMG respectively on the data collection form. Two observers blinded to the rest of the study and not involved with carrying out NCS / EMG will be trained to administer these scores. The guardian, who would be unaware of what the child scored, will also be shown the FPS-R and asked to score how much pain patient seemed to feel during NCS and EMG respectively. Regarding FPS-R, the instruction will be to choose the face that most closely resembles the amount of pain being felt. Patient demographics, Clinical characteristics and NCS / EMG procedure characteristics will also be recorded on the form. The data collected will then be entered into an excel sheet at the end of each day.

Sample Size:

Assuming a difference in means of 1.4 with a standard deviation of 1.73 in the control group and 2.17 in the intervention group on the MBPS according to a study assessing effectiveness of EMLA cream for reducing pain during Intramuscular injections in the pediatric population, an alpha level of 0.05 and power of 80 % using a 1-way analysis of variance (ANOVA) test with 3 pairwise comparisons; we will require 35 patients per group. Furthermore, assuming a 10 % dropout rate we will enroll 39 patients per group to account for it.

Randomization:

To achieve comparable groups, randomization will be performed as stratified blocked randomization with random sizes in a 1:1 allocation ratio. Stratification will be done according to the age groups: 6 months - 6 years and 7 - 18 years with varying random block sizes. Allocation to intervention groups according to stratification will be carried out by a computer generated randomization schedule which will list the allocation sequences assigned to each of the three arms. The randomization schedule will only be available with the pharmacist in charge of preparing interventions. Interventions will be prepared in indistinguishable containers containing plain cream and EMLA cream and bottles containing plain syrup and Ibuprofen syrup. The creams will be prepared to be similar in consistency, texture and color. The syrups will also be similar in color and taste. Thirty Nine Intervention packages will be made for each of the intervention arms; COTA arm, OA arm and Placebo arm. Each intervention will be labelled with an allocation sequence according to the randomization schedule by the pharmacist. The independent study officer not involved with the preparation or packaging of interventions and blinded to the rest of the study will issue the intervention for each patient reporting on the day of the appointment. The random allocation sequence would be concealed from the rest of the study investigators / researchers.

Blinding:

Throughout the study the patients, the electromyographers, neurophysiology technologists / observers administering the validated pain scales will be unaware of the intervention assignments.

Safety Management:

The drugs used in intervention arm have FDA approval as analgesics in the study population. Moreover, no prior testing is recommended before administration of these over the counter analgesics. Our study involves a single time use of these drugs only. Possible side effects (1-10%) with Ibuprofen include dizziness, epigastric pain, heart burn, nausea, rash, vomiting and renal failure (<1%). Possible side effects (>10%) with EMLA application include application site pallor/blanching, erythema/pain and application site oedema (1-10%), itching. Rare adverse effects (<1%) include methemoglobinemia and myocardial dysfunction. Patients will be observed for 15 minutes post study for the development of any side effects. If any side effect is observed, patients would be referred to consult respective speciality as deemed appropriate, as per the severity of adverse event. The patient or his/her guardian will bear the expenses. This would be mentioned at the time of taking informed consent.

Data Handling & Storage:

All patient related data would be kept safe in the custody of designated study officer who would be part of the neurophysiology lab. Informed consent forms would be signed in a separate room.

Statistical Analysis:

Data will be assessed for normality. We will use descriptive statistics for patient demographics, clinical characteristics and NCS / EMG test characteristics, including measures of central tendency and dispersion. Comparisons between three groups on pain perception will be performed using ANOVA. Differences in proportions will be assessed using chi-square test or Fischer exact test where appropriate. Logistic and Linear regression models will be used to assess the effect of patient demographics, clinical characteristics and NCS / EMG test characteristics on patient pain reduction within and across intervention groups. All p-values will be two sided and considered as statistically significant if < 0.05. All analyses will be conducted by using the Statistical package for social science SPSS (Release 19.0, standard version, copyright © SPSS; 1989-02).

ELIGIBILITY:
Inclusion Criteria:

- Pediatric patients (6 months to 18 years) referred for NCS / EMG testing to the neurophysiology lab at AKUH

Exclusion Criteria:

* Patients not able to report pain scores on the scales used
* Patients using sedatives and prior analgesics within last 24 hours of study
* Patients with history of upper gastrointestinal tract bleed, renal disease, severe hepatic disease, glucose-6-phosphate deficiency, congenital or idiopathic methemoglobinemia
* Patients with known sensitivity / allergy to Ibuprofen or EMLA cream or their components
* Patients on class I antiarrhythmic drugs
* Patients with breach of skin on topical analgesic/placebo application sites
* Breastfeeding or sugary drink within one hour of start of study

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 113 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Pain perception of patient during NCS and EMG tests | Pain scores to be recorded immediately after the procedure
  Pain perception of patient during NCS and EMG tests as measured by Modified Behavioral Pain Scale or patient reported Faces Pain Scale - Revised in COTA, OA and Placebo arms.

SECONDARY OUTCOMES:
Pain perception of patient according to guardian during NCS and EMG tests | Pain scores to be recorded immediately after the procedure
  Pain perception of patient according to guardian during NCS and EMG tests as measured by guardian-reported FPS-R
Effect of Patient demographics, Clinical characteristics and NCS / EMG procedure characteristics on patient pain scores | Pain scores to be recorded immediately after the procedure
  Effect of Patient demographics, Clinical characteristics and NCS / EMG procedure characteristics on patient pain scores within and across each of the intervention arms

CONTACTS AND LOCATIONS:
Overall Officials: Fazal Rehman, MBBS, FCPS, Principal Investigator — Aga Khan University; Haris Hakeem, MBBS, FCPS, FRACP, Principal Investigator — Aga Khan University Hospital, Monash University
Locations (1):
- Aga khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gans BM, Kraft GH. Pain perception in clinical electromyography. Arch Phys Med Rehabil. 1977 Jan;58(1):13-6. PMID 831658
- [Background] Strommen JA, Daube JR. Determinants of pain in needle electromyography. Clin Neurophysiol. 2001 Aug;112(8):1414-8. doi: 10.1016/s1388-2457(01)00552-1. PMID 11459681
- [Background] London ZN, Burke JF, Hazan R, Hastings MM, Callaghan BC. Electromyography-related pain: muscle selection is the key modifiable study characteristic. Muscle Nerve. 2014 Apr;49(4):570-4. doi: 10.1002/mus.23974. Epub 2014 Jan 25. PMID 23893537
- [Background] Yalinay Dikmen P, Ilgaz Aydinlar E, Karlikaya G. Expected and Experienced Pain Levels in Electromyography. Noro Psikiyatr Ars. 2013 Dec;50(4):364-367. doi: 10.4274/npa.y6699. Epub 2013 Dec 1. PMID 28360571
- [Background] Pohl M, Rosler A, Sunkeler I, Braune HJ, Oertel WH, Lautenbacher S. Insertion pain in needle electromyography can be reduced by simultaneous finger slapping. Neurology. 2000 Mar 14;54(5):1201-2. doi: 10.1212/wnl.54.5.1201-a. No abstract available. PMID 10720303
- [Background] Annaswamy TM, Morchower AH. Effect of lidocaine iontophoresis on pain during needle electromyography. Am J Phys Med Rehabil. 2011 Dec;90(12):961-8. doi: 10.1097/PHM.0b013e318228c6d3. PMID 22019960
- [Background] Lamarche Y, Lebel M, Martin R. EMLA partially relieves the pain of EMG needling. Can J Anaesth. 1992 Oct;39(8):805-8. doi: 10.1007/BF03008292. PMID 1288906
- [Background] Kalantar SS, Abbasi M, Faghihi-Kashani S, Majedi H, Ahmadi M, Agah E, Tafakhori A. Paracetamol 325 mg/tramadol 37.5 mg effect on pain during needle electromyography: a double-blind crossover clinical trial. Acta Neurol Belg. 2016 Dec;116(4):599-604. doi: 10.1007/s13760-016-0621-6. Epub 2016 Mar 8. PMID 26957290
- [Background] El-Salem K, Shakhatreh M. Prospective double-blind crossover trial of ibuprofen in reducing EMG pain. Muscle Nerve. 2008 Aug;38(2):1016-20. doi: 10.1002/mus.21017. PMID 18663736
- [Background] Alshaikh NM, Martinez JP, Pitt MC. Perception of pain during electromyography in children: A prospective study. Muscle Nerve. 2016 Sep;54(3):422-6. doi: 10.1002/mus.25069. Epub 2016 Feb 26. PMID 26852012
- [Background] Taddio A, Ilersich AL, Ipp M, Kikuta A, Shah V; HELPinKIDS Team. Physical interventions and injection techniques for reducing injection pain during routine childhood immunizations: systematic review of randomized controlled trials and quasi-randomized controlled trials. Clin Ther. 2009;31 Suppl 2:S48-76. doi: 10.1016/j.clinthera.2009.07.024. PMID 19781436
- [Background] Taddio A, Appleton M, Bortolussi R, Chambers C, Dubey V, Halperin S, Hanrahan A, Ipp M, Lockett D, MacDonald N, Midmer D, Mousmanis P, Palda V, Pielak K, Riddell RP, Rieder M, Scott J, Shah V. Reducing the pain of childhood vaccination: an evidence-based clinical practice guideline. CMAJ. 2010 Dec 14;182(18):E843-55. doi: 10.1503/cmaj.101720. Epub 2010 Nov 22. No abstract available. PMID 21098062
- [Background] Taddio A, Hogan ME, Moyer P, Girgis A, Gerges S, Wang L, Ipp M. Evaluation of the reliability, validity and practicality of 3 measures of acute pain in infants undergoing immunization injections. Vaccine. 2011 Feb 4;29(7):1390-4. doi: 10.1016/j.vaccine.2010.12.051. Epub 2010 Dec 30. PMID 21195076
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] von Baeyer CL. Children's self-reports of pain intensity: scale selection, limitations and interpretation. Pain Res Manag. 2006 Autumn;11(3):157-62. doi: 10.1155/2006/197616. PMID 16960632
- [Background] Abuelkheir M, Alsourani D, Al-Eyadhy A, Temsah MH, Meo SA, Alzamil F. EMLA(R) cream: a pain-relieving strategy for childhood vaccination. J Int Med Res. 2014 Apr;42(2):329-36. doi: 10.1177/0300060513509473. Epub 2014 Feb 5. PMID 24501164